CLINICAL TRIAL: NCT00415688
Title: A Randomized, Controlled Trial of a Low-Carbohydrate, Ketogenic Diet Versus a Low-Glycemic Index Diet for Obesity-Related Type 2 Diabetes
Brief Title: Lifestyle Modification for Obesity-Related Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Robert C. Atkins Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF001
Record Dates: First submitted 2006-12-21; First posted 2006-12-25 (Estimated); Last update posted 2006-12-25 (Estimated); Status verified 2006-12

CONDITIONS: Type 2 Diabetes Mellitus; Overweight; Obesity
Keywords: lifestyle modification; weight loss; hyperglycemia; hypoglycemic agents
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Weight Loss; Hyperglycemia | interventions — Diet, Ketogenic

INTERVENTIONS:
Behavioral: Low carbohydrate, ketogenic diet
Behavioral: Low glycemic index, reduced calorie diet

SUMMARY:
Dietary carbohydrate is the major determinant of postprandial glucose levels, and preliminary evidence suggests that low carbohydrate diets improve glycemic control when accompanied by weight loss. To determine if glycemic control can be improved by varying dietary carbohydrate during weight loss, we compared two weight loss diets with different carbohydrate levels for the treatment of obesity-related type 2 diabetes over 24 weeks in the outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus for at least one year
* hgba1c > 6.0
* BMI from 27-50 kg/m2

Exclusion Criteria:

* Unstable medical condition
* Serious medical condition
* AST or ALT > 100
* Serum creatinine > 1.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2004-07; Study Completion 2006-01

PRIMARY OUTCOMES:
Hemoglobin A1c

SECONDARY OUTCOMES:
Body weight
Serum lipoproteins

CONTACTS AND LOCATIONS:
Overall Officials: Eric C Westman, MD MHS, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States